CLINICAL TRIAL: NCT03760458
Title: Phase I/II Study of the Pharmacokinetics, Safety, and Tolerability of Abacavir/Dolutegravir/Lamivudine Dispersible and Immediate Release Tablets in HIV-1-Infected Children Less Than 12 Years of Age
Brief Title: The Pharmacokinetics, Safety, and Tolerability of Abacavir/Dolutegravir/Lamivudine Dispersible and Immediate Release Tablets in HIV-1-Infected Children Less Than 12 Years of Age
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Mental Health (NIMH) (NIH); ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPAACT 2019; 38504 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-11-29; First posted 2018-11-30 (Actual); Results first posted 2023-02-13 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-05

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — abacavir; abacavir, dolutegravir, and lamivudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Weight Band #1 (6 to less than 10 kg at study entry) (Experimental): Children weighing 6 to less than 10 kg at study entry. These children received 3 dispersible tablets of ABC/DTG/3TC daily while weighing 6-<10 kg; as their weight increased, they received higher doses consistent with their new weight band.
  Interventions: Drug: Abacavir (ABC)/Dolutegravir (DTG)/Lamivudine (3TC) Dispersible Tablets
- Weight Band #2 (10 to less than 14 kg at study entry) (Experimental): Children weighing 10 to less than 14 kg at study entry. These children received 4 dispersible tablets of ABC/DTG/3TC daily while weighing 10-<14 kg; as their weight increased, they received higher doses consistent with their new weight band.
  Interventions: Drug: Abacavir (ABC)/Dolutegravir (DTG)/Lamivudine (3TC) Dispersible Tablets
- Weight Band #3 (14 to less than 20 kg at study entry) (Experimental): Children weighing 14 to less than 20 kg at study entry. These children received 5 dispersible tablets of ABC/DTG/3TC daily while weighing 14-<20 kg; as their weight increased, they received higher doses consistent with their new weight band.
  Interventions: Drug: Abacavir (ABC)/Dolutegravir (DTG)/Lamivudine (3TC) Dispersible Tablets
- Weight Band #4 (20 to less than 25 kg at study entry) (Experimental): Children weighing 20 to less than 25 kg at study entry. These children received 6 dispersible tablets of ABC/DTG/3TC daily while weighing 20-<25 kg; as their weight increased, they received higher doses consistent with their new weight band.
  Interventions: Drug: Abacavir (ABC)/Dolutegravir (DTG)/Lamivudine (3TC) Dispersible Tablets
- Weight Band #5 (25 kg or greater at study entry) (Experimental): Children weighing 25 kg or greater at study entry. These children received 1 immediate release tablet of ABC/DTG/3TC daily.
  Interventions: Drug: Abacavir (ABC)/Dolutegravir (DTG)/Lamivudine (3TC) Immediate Release Tablets (Immediate release)

INTERVENTIONS:
Drug: Abacavir (ABC)/Dolutegravir (DTG)/Lamivudine (3TC) Dispersible Tablets — Fixed-dose combination dispersible tablets containing 60 mg ABC, 5 mg DTG, and 30 mg 3TC; administered orally once daily with or without food
  Arms: Weight Band #1 (6 to less than 10 kg at study entry); Weight Band #2 (10 to less than 14 kg at study entry); Weight Band #3 (14 to less than 20 kg at study entry); Weight Band #4 (20 to less than 25 kg at study entry)
Drug: Abacavir (ABC)/Dolutegravir (DTG)/Lamivudine (3TC) Immediate Release Tablets (Immediate release) — Fixed-dose combination immediate release tablets containing 600 mg ABC, 50 mg DTG, and 300 mg 3TC; administered orally once daily with or without food
  Other Names: Triumeq
  Arms: Weight Band #5 (25 kg or greater at study entry)

SUMMARY:
The purpose of this study was to examine the pharmacokinetics, safety, and tolerability of abacavir/dolutegravir/lamivudine dispersible and immediate release tablets in children living with HIV less than 12 years of age.

DETAILED DESCRIPTION:
This study examined the pharmacokinetics (PK), safety, and tolerability of fixed-dose combination abacavir (ABC)/dolutegravir (DTG)/lamivudine (3TC) dispersible and immediate release tablets in children living with HIV less than 12 years of age.

Children were enrolled into one of five ABC/DTG/3TC dosing groups based on their weight. The first 5-7 children within each weight-band underwent intensive PK assessments 5-10 days after starting ABC/DTG/3TC to confirm dose selection. Children remained on their initial dose of ABC/DTG/3TC through Week 4. After Week 4, ABC/DTG/3TC dosing was adjusted based on PK results at the individual or weight-band level, and/or an individual child's growth and weight gain over time.

Follow-up study visits for all participants occurred at Weeks 1, 4, 12, 24, 36, and 48. If participants had a known M184 resistance mutation, they had additional study visits at Weeks 8, 16, and 20. Study visits included physical examination, study drug adherence and tolerability questionnaires, blood collection, and intensive PK sampling. Following the Week 48 study visit, some children were allowed to continue follow-up through up to 144 weeks if alternative post-study drug supply was not yet available.

ELIGIBILITY:
Inclusion Criteria:

* Weight 6 kg to less than 40 kg at entry
* Antiretroviral therapy (ART)-naïve at entry or has been taking a stable ART regimen for at least six consecutive months at entry

  * Note: For ART-naïve children, receipt of antiretroviral (ARV) prophylaxis prior to diagnosis of HIV infection is permitted. For these children, ascertainment of this criterion may be based on parent or guardian report only, but available medical records should also be reviewed in relation to this criterion.
  * Note: For ART-experienced children (on a stable ART regimen), dose and formulation changes (e.g., for growth) within the six months prior to entry are permitted. For these children, ascertainment of this criterion must be based on medical records.
* For ART-experienced children (on a stable ART regimen), has had a suppressed HIV viral load (HIV-1 RNA less than 200 copies/mL) for at least six consecutive months prior to entry

  * Note: To fulfill this criterion, at least two documented HIV-1 RNA results less than 200 copies/mL must be available, one based on a specimen collected at least six months prior to entry and one based on a specimen collected within 30 days prior to entry.
  * Note: Any documented HIV-1 RNA result greater than or equal to 200 copies/mL based on a specimen collected within six months prior to entry is exclusionary (see exclusion criterion below).
* At screening, has normal, Grade 1, or Grade 2 laboratory test results for all of the following, based on testing of specimens collected within 30 days prior to entry and grading per the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (refer to the study protocol for guidance on severity grading):

  * Hemoglobin (greater than or equal to 8.5 g/dL or greater than or equal to 5.25 mmol/L)
  * Absolute neutrophil count (greater than or equal to 600 cells/mm^3 or greater than or equal to 0.600 x 10^9 cells/L)
  * Platelet count (greater than or equal to 50,000 cells/mm^3 or greater than or equal to 50.00 x 10^9 cells/L)
  * Estimated glomerular filtration rate (eGFR; bedside Schwartz formula; greater than or equal to 60 ml/min/1.73 m^2)
  * Alanine transaminase (ALT) (less than 5.0 x ULN)
  * Aspartate aminotransferase (AST) (less than 5.0 x ULN)
  * Total bilirubin (less than 2.6 x ULN)
  * Direct bilirubin (less than or equal to ULN)
  * Note: Laboratory tests may be repeated during the screening period (i.e., within 30 days prior to entry), with the latest results used for eligibility determination.
  * Note: For treatment-experienced children on an atazanavir-containing ART regimen, Grade 3 or higher total bilirubin is permitted.
* At screening, has a negative test result for hepatitis B surface antigen based on testing of a specimen collected within 30 days prior to entry
* Confirmed HIV-1-infection based on documented testing of two samples collected at different time points:

  * Sample #1 may be tested using any of the following:

    * Two rapid antibody tests from different manufacturers or based on different principles and epitopes
    * One enzyme immunoassay OR Western Blot OR immunofluorescence assay OR chemiluminescence assay
    * One HIV DNA polymerase chain reaction (PCR)*
    * One quantitative HIV RNA PCR (above the limit of detection of the assay)*
    * One qualitative HIV RNA PCR*
    * One HIV total nucleic acid test*
  * Sample #2 may be tested using any of the following:

    * Rapid antibody test. If this option is used in combination with two rapid tests for Sample #1, at least one of the three rapid tests must be United States Food and Drug Administration (FDA)-approved, and the third rapid test must be from a third manufacturer or based on a third principle or epitope.
    * One enzyme immunoassay OR Western Blot OR immunofluorescence assay OR chemiluminescence assay
    * One HIV DNA PCR*
    * One quantitative HIV RNA PCR (above the limit of detection of the assay)*
    * One qualitative HIV RNA PCR*
    * One HIV total nucleic acid test*
  * For participants who are less than two years of age, or who are two years of age and older with any exposure to breast milk in the past 28 days, HIV-1 infection must be confirmed using the tests indicated above with an asterisk (*) for Sample #1 and Sample #2.
  * Whole blood, plasma, or serum samples must be tested. If both samples are tested using antibody tests, at least one of the samples must be tested in a laboratory that operates according to Good Clinical Laboratory Practice guidelines and participates in an appropriate external quality assurance program. If nucleic acid testing is used, at least one test must be performed in a Clinical Laboratory Improvement Amendments (CLIA) certified (for US sites) or Virology Quality Assurance (VQA) certified (for non-US sites) laboratory. For tests performed in other settings, adequate source documentation including the date of specimen collection, date of testing, test performed, and test result must be available. FDA approved testing methods should be used when possible.
* HLA-B*5701-negative based on documented testing at any time prior to entry

  * Note: Documented testing is required even if the potential participant has received ABC prior to study entry.
* For females of reproductive potential (defined as having experienced menarche), not pregnant based on testing performed at screening
* For females of reproductive potential who are engaging in sexual activity that could lead to pregnancy, willing to use two methods of contraception while receiving study drug, based on participant and parent or guardian report at entry

  * One of the two methods must be highly effective; highly effective methods include surgical sterilization (i.e., hysterectomy, bilateral oophorectomy, tubal ligation, or salpingectomy) and the following:

    * Contraceptive intrauterine device or intrauterine system
    * Subdermal contraceptive implant
    * Progestogen injections
    * Combined estrogen and progestogen oral contraceptive pills
    * Percutaneous contraceptive patch
    * Contraceptive vaginal ring
  * The highly effective method must be initiated prior to study entry. The second method should ideally be a barrier method. Male or female condom use is recommended with all other methods of contraception for dual protection against pregnancy and to avoid transmission of HIV and other sexually transmitted infections.
* Based on parent or guardian report at entry, child is expected to be available for 48 weeks of follow-up
* Parent or legal guardian is willing and able to provide written informed consent for child's study participation and, when applicable per local institutional review board/ethics committee (IRB/EC) policies and procedures, child is willing and able to provide written informed assent for study participation

Exclusion Criteria:

* Documented resistance to ABC, DTG, or 3TC

  * Note: Testing to rule out resistance is not required, and the M184V resistance mutation is not exclusionary.
* For ART-experienced children (on a stable ART regimen), documented HIV-1 RNA result greater than or equal to 200 copies/mL based on a specimen collected within six months prior to entry
* History of any of the following as determined by the site investigator based on participant/parent/guardian report and available medical records:

  * Malignancy (ever)
  * Hypersensitivity reaction to ABC (ever)
  * Receipt of any prohibited medication (refer to the study protocol for more information) within 30 days prior to study entry
  * Receipt of systemic interferon or any chronic systemic immunosuppressant medication within 30 days prior to study entry
  * Note: Systemic corticosteroids (e.g., prednisone or equivalent up to 2 mg/kg) taken for replacement or short course therapy are permitted. Intranasal or inhaled steroid use is also permitted.
* Has any of the following as determined by the site investigator based on participant/parent/guardian report and available medical records

  * Current clinical evidence of pancreatitis
  * Currently-active tuberculosis (TB) and/or currently receiving rifampicin-containing TB treatment
  * Currently-active AIDS-defining (WHO Clinical Stage 4) opportunistic infection
* Has any documented or suspected clinically significant medical condition or any other condition that, in the opinion of the site investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Flynn, MD, Study Chair — St. Jude Children's Research Hospital; Helena Rabie, MBChB, MMED, FCPaed, Study Chair — University of Stellenbosch; Jennifer Kiser, PharmD, PhD, Study Chair — University of Colorado Skaggs School of Pharmacy and Pharmaceutical Sciences
Locations (14):
- United States (5):
  - David Geffen School of Medicine at UCLA NICHD CRS, Los Angeles, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Rush Univ. Cook County Hosp. Chicago NICHD CRS, Chicago, Illinois
  - Lurie Children's Hospital of Chicago (LCH) CRS, Chicago, Illinois
  - St. Jude Children's Research Hospital CRS, Memphis, Tennessee
- Botswana (2):
  - Gaborone CRS, Gaborone
  - Molepolole CRS, Gaborone
- South Africa (4):
  - Soweto IMPAACT CRS, Johannesburg, Gauteng
  - Wits RHI Shandukani Research Centre CRS, Johannesburg, Gauteng
  - Umlazi CRS, Umlazi, KwaZulu-Natal
  - Famcru Crs, Tygerberg, Western Cape
- Thailand (3):
  - Siriraj Hospital, Mahidol University NICHD CRS, Bangkok, Bangkoknoi
  - Chiangrai Prachanukroh Hospital NICHD CRS, Changklan, Muang, Chiang Mai
  - Chiang Mai University HIV Treatment (CMU HIV Treatment) CRS, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom?
    * Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses?
    * To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available?
    * Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/studies/submit-research-proposal. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.

REFERENCES:
- [Derived] Brooks KM, Kiser JJ, Ziemba L, Ward S, Rani Y, Cressey TR, Masheto GR, Cassim H, Deville JG, Ponatshego PL, Patel F, Aurpibul L, Barnabas SL, Mustich I, Coletti A, Heckman B, Krotje C, Lojacono M, Yin DE, Townley E, Moye J, Majji S, Acosta EP, Ryan K, Chandasana H, Brothers CH, Buchanan AM, Rabie H, Flynn PM; IMPAACT 2019 Study Team. Pharmacokinetics, safety, and tolerability of dispersible and immediate-release abacavir, dolutegravir, and lamivudine tablets in children with HIV (IMPAACT 2019): week 24 results of an open-label, multicentre, phase 1-2 dose-confirmation study. Lancet HIV. 2023 Aug;10(8):e506-e517. doi: 10.1016/S2352-3018(23)00107-8. PMID 37541705
- [Derived] Singh RP, Adkison KK, Baker M, Parasrampuria R, Wolstenholme A, Davies M, Sewell N, Brothers C, Buchanan AM. Development of Dolutegravir Single-entity and Fixed-dose Combination Formulations for Children. Pediatr Infect Dis J. 2022 Mar 1;41(3):230-237. doi: 10.1097/INF.0000000000003366. PMID 34817414
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1 (July 2017) — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual), Version 2.0, January 2010 — http://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids
- See also: FDA Snapshot Algorithm — https://www.fda.gov/files/drugs/published/Human-Immunodeficiency-Virus-1-Infection--Developing-Antiretroviral-Drugs-for-Treatment.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual occurred between September 2020 and June 2021 in Botswana, South Africa, Thailand, and the United States at 14 different medical clinic sites.
Period: Main Study (Through Week 48)
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Started | 9 | 12 | 15 | 10 | 11
Completed | 8 | 11 | 15 | 10 | 11
Not Completed | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Period: Extended Follow-up (Weeks 48 Through 60)
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Started | 0 | 0 | 4 | 3 | 3
Completed | 0 | 0 | 4 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry) | Total
Number analyzed (Participants) | 9 | 12 | 15 | 10 | 11 | 57
Age, Continuous [Median (Full Range); unit: years] | 1.35 [0.98 to 2.02] | 3.56 [1.51 to 4.51] | 6.44 [3.88 to 9.58] | 8.41 [6.38 to 8.91] | 9.74 [8.68 to 11.28] | 6.38 [0.98 to 11.28]
Age, Customized [Count of Participants; unit: Participants]
  <6 years | 9 | 12 | 7 | 0 | 0 | 28
  6 to <12 years | 0 | 0 | 8 | 10 | 11 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 5 | 3 | 6 | 26
  Male | 4 | 5 | 10 | 7 | 5 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 3 | 3
  Not Hispanic or Latino | 9 | 12 | 15 | 10 | 7 | 53
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 1 | 7 | 4 | 3 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 10 | 7 | 6 | 8 | 37
  White | 0 | 1 | 0 | 0 | 0 | 1
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 0 | 2 | 2 | 1 | 5 | 10
  Botswana | 4 | 2 | 3 | 2 | 2 | 13
  South Africa | 2 | 7 | 4 | 3 | 1 | 17
  Thailand | 3 | 1 | 6 | 4 | 3 | 17
Weight [Median (Inter-Quartile Range); unit: kilograms] | 9.2 [8.5 to 9.5] | 12.9 [12.5 to 13.7] | 17.0 [15.9 to 18.8] | 21.5 [21.0 to 23.3] | 28.5 [26.0 to 35.6] | 17.0 [12.8 to 22.1]
Pre-study Antiretroviral (ART) experience [Count of Participants; unit: Participants]
  ART-experienced | 6 | 12 | 15 | 10 | 11 | 54
  ART-naive | 3 | 0 | 0 | 0 | 0 | 3
Known M184V mutation [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 2 | 0 | 2 | 4
  No | 9 | 12 | 13 | 10 | 9 | 53
HIV-1 RNA [Count of Participants; unit: Participants] — Viral loads less than the lower limit of quantification were imputed as one less than the lower limit.
  Participants
    <200 copies/mL | 5 | 12 | 15 | 10 | 11 | 53
    ≥200 copies/mL | 4 | 0 | 0 | 0 | 0 | 4
CD4+ Cell Count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: CD4 was not collected at baseline for one participant in Weight Band #2.
  cells/mm^3
    number analyzed (Participants) | 9 | 11 | 15 | 10 | 11 | 56
    (all) | 2321 [1390 to 3514] | 1452 [1161 to 2615] | 886 [761 to 1412] | 1155 [801 to 1251] | 915 [753 to 1450] | 1201 [880 to 1535]
CD4+ Percentage [Median (Inter-Quartile Range); unit: percentage of CD4+ in total lymphocytes] — Population: CD4/Lymphocytes was not collected at baseline for one participant in Weight Band #2.
  percentage of CD4+ in total lymphocytes
    number analyzed (Participants) | 9 | 11 | 15 | 10 | 11 | 56
    (all) | 34.0 [32.3 to 49.1] | 33.9 [31.6 to 45.6] | 32.9 [31.6 to 39.2] | 32.6 [26.2 to 43.0] | 37.7 [35.6 to 43.0] | 35.1 [31.9 to 43.0]
Total Cholesterol [Median (Inter-Quartile Range); unit: mmol/L] | 4.01 [3.19 to 4.82] | 4.61 [3.39 to 5.11] | 4.51 [3.70 to 5.20] | 5.19 [3.86 to 5.90] | 4.27 [3.25 to 5.72] | 4.51 [3.57 to 5.30]
High-Density Lipoprotein (HDL) Cholesterol [Median (Inter-Quartile Range); unit: mmol/L] | 0.98 [0.96 to 1.18] | 1.53 [1.29 to 1.63] | 1.38 [1.24 to 1.79] | 1.67 [1.14 to 2.00] | 1.34 [1.13 to 1.53] | 1.37 [1.1914 to 1.67]
Low-Density Lipoprotein (LDL) Cholesterol [Median (Inter-Quartile Range); unit: mmol/L] | 2.52 [1.92 to 3.20] | 2.25 [2.00 to 3.01] | 2.50 [1.94 to 3.03] | 3.04 [2.31 to 3.55] | 2.36 [1.79 to 3.09] | 2.52 [1.93 to 3.10]
Triglycerides [Median (Inter-Quartile Range); unit: mmol/L] | 1.71 [1.04 to 2.00] | 1.20 [0.94 to 1.75] | 1.23 [0.90 to 1.57] | 1.08 [0.81 to 1.32] | 1.76 [0.75 to 2.88] | 1.20 [0.90 to 1.76]

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Area Under the Plasma Concentration-time Curve Over 24 Hours (AUC0-24h) for ABC, DTG, and 3TC
Description: Based on analysis of intensive pharmacokinetic (PK) samples. The geometric mean AUC0-24h for each Weight Band was compared to the lower and upper reference values (in ug*h/mL) for DTG (35.1, 134), ABC (6.3, 50.4), and 3TC (6.3, 26.5). Steady state was measured at Week 1, but was re-collected later for two participants due to a specimen handling error for the Week 1 specimens.
Time Frame: Week 1; Blood samples were drawn at pre-dose and 1, 2, 3, 4, 6, 8, and 24 hours post dosing.
Population: Participants receiving treatment at timepoint who received treatment for their enrollment weight band through the intensive PK collection, and through either the Week 4 visit or the occurrence of an adverse event prior to the Week 4 visit that 1) was grade 3 or higher and assessed as related to study drug, or 2) resulted in premature discontinuation of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
h*ug/mL
  Abacavir (ABC) | 17.7 (33.8) | 19.8 (50.6) | 15.1 (40.3) | 17.4 (19.4) | 25.7 (14.6)
  Dolutegravir (DTG) | 75.9 (33.7) | 91.0 (36.5) | 71.4 (23.5) | 84.4 (26.3) | 71.8 (13.9)
  Lamivudine (3TC) | 10.7 (46.0) | 14.2 (23.9) | 13.0 (15.6) | 14.5 (16.6) | 21.7 (26.2)

2. Primary Outcome: Geometric Mean Maximum Plasma Concentration (Cmax) for ABC, DTG, and 3TC
Description: Based on analysis of intensive PK samples. Steady state was measured at Week 1, but was re-collected later for two participants due to a specimen handling error for the Week 1 specimens.
Time Frame: Week 1; Blood samples were drawn at pre-dose and 1, 2, 3, 4, 6, 8, and 24 hours post dosing.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
ug/mL
  ABC | 7.30 (20.5) | 8.36 (43.7) | 6.26 (31.0) | 6.65 (27.7) | 9.04 (21.9)
  DTG | 7.40 (28.0) | 8.85 (21.3) | 7.04 (17.0) | 7.29 (16.7) | 6.25 (20.6)
  3TC | 2.29 (39.8) | 3.55 (18.7) | 2.92 (23.0) | 2.99 (31.9) | 4.15 (29.3)

3. Primary Outcome: Geometric Mean Concentration at 24 Hours Post-dose (C24h) for ABC, DTG, and 3TC
Description: Based on analysis of intensive PK samples. The geometric mean C24h for each Weight Band was compared to the lower and upper reference values (in ug/mL) for DTG (0.67, 2.97). Steady state was measured at Week 1, but was re-collected later for two participants due to a specimen handling error for the Week 1 specimens.
Time Frame: Week 1; Blood samples were drawn at pre-dose and 1, 2, 3, 4, 6, 8, and 24 hours post dosing.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 7 | 7 | 7 | 7 | 7
ug/mL
  ABC | 0.003 (127.6) | 0.005 (127.4) | 0.003 (107.5) | 0.004 (84.9) | 0.011 (228.5)
  DTG | 0.91 (67.6) | 1.22 (77.5) | 0.79 (44.2) | 1.35 (95.5) | 0.98 (27.9)
  3TC | 0.055 (39.5) | 0.046 (48.3) | 0.058 (36.7) | 0.060 (18.3) | 0.084 (35.0)

4. Primary Outcome: Percentage of Participants Who Had at Least One Adverse Event Through Week 24
Description: Adverse event (AE) grading was based on the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Corrected Version 2.1, dated July 2017. AEs of any grade were reported.
Time Frame: Measured from treatment initiation through Week 24
Population: All participants who started treatment for their enrollment weight band and whose dose may have been increased to a higher weight band due to weight gain, who either completed treatment through Week 24 or discontinued treatment due to toxicity prior to Week 24.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 100.0 [63.1 to 100.0] | 90.9 [58.7 to 99.8] | 100.0 [78.2 to 100.0] | 80.0 [44.4 to 97.5] | 80.0 [44.4 to 97.5]

5. Primary Outcome: Percentage of Participants Who Had at Least One Grade 3 or Grade 4 Adverse Event Assessed as Related to Study Drug Through Week 24
Description: AE grading was based on DAIDS AE Grading Table, Corrected Version 2.1, dated July 2017. AEs of any grade were reported. The relationship to study drug was assessed by the site investigator.
Time Frame: Measured from treatment initiation through Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

6. Primary Outcome: Percentage of Participants Who Had a Grade 5 Adverse Event Assessed as Related to Study Drug Through Week 24
Description: as for outcome 5
Time Frame: Measured from treatment initiation through Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

7. Primary Outcome: Percentage of Participants Who Had at Least One Life-threatening Adverse Event Assessed as Related to Study Drug Through Week 24
Description: AE grading was based on DAIDS AE Grading Table, Corrected Version 2.1, dated July 2017. AEs of any grade were reported. The relationship to study drug was assessed by the site investigator. Life-threatening was defined according to Version 2.0 of the Manual for Expedited Reporting of Adverse Events to DAIDS (DAIDS EAE Manual).
Time Frame: Measured from treatment initiation through Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

8. Primary Outcome: Percentage of Participants Who Had at Least One Serious Adverse Event Assessed as Related to Study Drug Through Week 24
Description: AE grading was based on DAIDS AE Grading Table, Corrected Version 2.1, dated July 2017. AEs of any grade were reported. The relationship to study drug was assessed by the site investigator. Seriousness was defined according to Version 2.0 of the DAIDS EAE Manual.
Time Frame: Measured from treatment initiation through Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

9. Primary Outcome: Percentage of Participants Who Had at Least One Adverse Event Assessed as Related to Study Drug That Led to Permanent Discontinuation of Study Drug Through Week 24
Description: as for outcome 5
Time Frame: Measured from treatment initiation through Week 24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

10. Secondary Outcome: Population PK: Geometric Mean AUC0-24h for ABC, DTG, and 3TC
Description: Population PK: Geometric Mean Area Under the Plasma Concentration-time Curve for ABC, DTG, and 3TC derived from population PK model. Population apparent oral clearance and apparent volume of distribution were determined with non-linear mixed effects modeling. DTG and 3TC were fit to a 1-compartment model and ABC was fit to 2-compartment model. Weight was a covariate on clearance and volume for all drugs and enzyme maturation as a covariate on apparent oral clearance for DTG. The posthoc parameter of AUC0-24 was estimated using non-compartmental analysis of simulated steady-state concentration-time profiles and stratified by weight band.
Time Frame: Measured from Week 1 through Week 48 over 24 hours post-dose
Population: All participants with intensive or sparse PK results at the recommended doses according to their enrollment weight band. Two participants who discontinued the study in the first week were not included
Measure: Geometric Mean (95% Confidence Interval); unit: ug*h/mL
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
ug*h/mL
  ABC | 17.30 [12 to 25.1] | 18.90 [14.7 to 24.2] | 17.20 [14.8 to 20] | 19.50 [16.6 to 22.9] | 26.10 [22.5 to 30.2]
  DTG | 82.20 [65.6 to 103] | 86.90 [75.3 to 100] | 71.50 [62.1 to 82.2] | 81.60 [70.8 to 94.2] | 72.60 [64.9 to 81.1]
  3TC | 9.97 [7.12 to 14] | 14.90 [10.6 to 20.9] | 13.60 [11.6 to 15.8] | 13.10 [11.2 to 15.2] | 20.30 [16.9 to 24.3]

11. Secondary Outcome: Population PK: Geometric Mean Concentration at Time 0 (Pre-dose) (C0h) for ABC, DTG, and 3TC
Description: as for outcome 10
Time Frame: Measured from Week 1 through Week 48 over 24 hours post-dose
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
ug/mL
  ABC | 0.01 [0.002 to 0.021] | 0.02 [0.007 to 0.042] | 0.01 [0.008 to 0.021] | 0.01 [0.004 to 0.015] | 0.02 [0.010 to 0.038]
  DTG | 1.08 [0.67 to 1.74] | 1.35 [1.01 to 1.82] | 0.71 [0.478 to 1.05] | 1.09 [0.761 to 1.56] | 1.01 [0.772 to 1.32]
  3TC | 0.01 [0.003 to 0.015] | 0.03 [0.01 to 0.085] | 0.02 [0.006 to 0.04] | 0.01 [0.003 to 0.028] | 0.02 [0.008 to 0.074]

12. Secondary Outcome: Population PK: Geometric Mean Concentration at 24 Hours Post-dose (C24h) for ABC, DTG, and 3TC
Description: as for outcome 10
Time Frame: Measured from Week 1 through Week 48 over 24 hours post-dose
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
ug/mL
  ABC | 0.01 [0.003 to 0.018] | 0.02 [0.007 to 0.042] | 0.01 [0.007 to 0.024] | 0.01 [0.004 to 0.018] | 0.02 [0.010 to 0.040]
  DTG | 1.08 [0.67 to 1.74] | 1.35 [1.01 to 1.82] | 0.71 [0.48 to 1.05] | 1.09 [0.76 to 1.56] | 1.01 [0.77 to 1.32]
  3TC | 0.01 [0.004 to 0.047] | 0.02 [0.005 to 0.053] | 0.01 [0.005 to 0.021] | 0.02 [0.007 to 0.043] | 0.03 [0.008 to 0.081]

13. Secondary Outcome: Population PK: Geometric Mean Maximum Plasma Concentration (Cmax) for ABC, DTG, and 3TC
Description: as for outcome 10
Time Frame: Measured from Week 1 through Week 48 over 24 hours post-dose
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
ug/mL
  ABC | 6.04 [4.29 to 8.51] | 7.42 [5.75 to 9.57] | 7.07 [5.73 to 8.73] | 8.04 [6.27 to 10.3] | 9.60 [8.03 to 11.5]
  DTG | 6.79 [5.92 to 7.8] | 6.63 [5.96 to 7.37] | 6.36 [5.9 to 6.85] | 6.59 [6.13 to 7.09] | 5.43 [4.91 to 6.02]
  3TC | 2.29 [1.82 to 2.88] | 2.64 [2.12 to 3.29] | 2.98 [2.65 to 3.35] | 2.65 [2.16 to 3.25] | 3.59 [2.89 to 4.45]

14. Secondary Outcome: Population PK: Geometric Mean Time to Maximum Concentration (Tmax) for ABC, DTG, and 3TC
Description: as for outcome 10
Time Frame: Measured from Week 1 through Week 48 over 24 hours post-dose
Population: as for outcome 10
Measure: Median (Full Range); unit: hours
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
hours
  ABC | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00]
  DTG | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 4.00] | 2.00 [2.00 to 4.00] | 2.50 [1.00 to 4.00] | 3.00 [2.00 to 6.00]
  3TC | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 8.00] | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00] | 2.00 [2.00 to 4.00]

15. Secondary Outcome: Population PK: Geometric Mean Apparent Oral Clearance (CL/F) for ABC, DTG, and 3TC
Description: as for outcome 10
Time Frame: Measured from Week 1 through Week 48 over 24 hours post-dose
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: L/hour
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
L/hour
  ABC | 10.40 [7.16 to 15.1] | 12.70 [9.92 to 16.3] | 17.40 [15 to 20.2] | 18.40 [15.7 to 21.7] | 23.00 [19.8 to 26.6]
  DTG | 0.18 [0.15 to 0.23] | 0.23 [0.20 to 0.27] | 0.35 [0.30 to 0.40] | 0.37 [0.32 to 0.42] | 0.69 [0.62 to 0.77]
  3TC | 9.03 [6.45 to 12.6] | 8.04 [5.74 to 11.3] | 11.00 [9.46 to 12.9] | 13.80 [11.8 to 16] | 14.80 [12.3 to 17.7]

16. Secondary Outcome: Population PK: Geometric Mean Half-life (t1/2) for ABC, DTG, and 3TC
Description: as for outcome 10
Time Frame: Measured from Week 1 through Week 48 over 24 hours post-dose
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
hours
  ABC | 3.21 [2.54 to 4.07] | 3.43 [2.71 to 4.34] | 3.72 [3.19 to 4.33] | 3.32 [2.75 to 4.01] | 3.30 [2.75 to 3.97]
  DTG | 8.34 [6.68 to 10.4] | 9.42 [7.91 to 11.2] | 6.75 [5.82 to 7.83] | 8.34 [6.72 to 10.4] | 8.14 [7 to 9.46]
  3TC | 3.38 [2.54 to 4.48] | 3.23 [2.5 to 4.16] | 2.97 [2.52 to 3.49] | 3.46 [2.64 to 4.52] | 3.51 [2.64 to 4.66]

17. Secondary Outcome: Percentage of Participants With at Least One Adverse Event Through Week 48
Description: AE grading was based on DAIDS AE Grading Table, Corrected Version 2.1, dated July 2017. AEs of any grade were reported.
Time Frame: Measured from treatment initiation through Week 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 100.0 [63.1 to 100.0] | 90.9 [58.7 to 99.8] | 100.0 [78.2 to 100.0] | 100.0 [69.2 to 100.0] | 90.0 [55.5 to 99.7]

18. Secondary Outcome: Percentage of Participants Who Had at Least One Grade 3 or Grade 4 Adverse Event Assessed as Related to Study Drug Through Week 48
Description: as for outcome 5
Time Frame: Measured from treatment initiation through Week 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 20.0 [2.5 to 55.6] | 0.0 [0.0 to 30.8]

19. Secondary Outcome: Percentage of Participants Who Had a Grade 5 Adverse Event Assessed as Related to Study Drug Through Week 48
Description: as for outcome 5
Time Frame: Measured from treatment initiation through Week 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

20. Secondary Outcome: Percentage of Participants Who Had at Least One Life-threatening Adverse Event Assessed as Related to Study Drug Through Week 48
Description: AE grading was based on DAIDS AE Grading Table, Corrected Version 2.1, dated July 2017. AEs of any grade were reported. The relationship to study drug was assessed by the site investigator. Life-threatening was defined according to Version 2.0 of the DAIDS EAE Manual.
Time Frame: Measured from treatment initiation through Week 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

21. Secondary Outcome: Percentage of Participants Who Had at Least One Serious Adverse Event Assessed as Related to Study Drug Through Week 48
Description: as for outcome 8
Time Frame: Measured from treatment initiation through Week 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 30.8]

22. Secondary Outcome: Percentage of Participants Who Had at Least One Adverse Event Assessed as Related to Study Drug That Led to Permanent Discontinuation of Study Drug Through Week 48
Description: as for outcome 5
Time Frame: Measured from treatment initiation through Week 48
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 30.8]

23. Secondary Outcome: Percentage of Participants Who Had at Least One Adverse Event Through Week 60
Description: AE grading was based on DAIDS AE Grading Table, Corrected Version 2.1, dated July 2017. AEs of any grade were reported.
Time Frame: Measured from treatment initiation through Week 60
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 100.0 [63.1 to 100.0] | 90.9 [58.7 to 99.8] | 100.0 [78.2 to 100.0] | 100.0 [69.2 to 100.0] | 90.0 [55.5 to 99.7]

24. Secondary Outcome: Percentage of Participants Who Had at Least One Grade 3 or Grade 4 Adverse Event Assessed as Related to Study Drug Through Week 60
Description: as for outcome 5
Time Frame: Measured from treatment initiation through Week 60
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 20.0 [2.5 to 55.6] | 0.0 [0.0 to 30.8]

25. Secondary Outcome: Percentage of Participants Who Had a Grade 5 Adverse Event Assessed as Related to Study Drug Through Week 60
Description: as for outcome 5
Time Frame: Measured from treatment initiation through Week 60
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

26. Secondary Outcome: Percentage of Participants Who Had at Least One Life-threatening Adverse Event Assessed as Related to Study Drug Through Week 60
Description: as for outcome 20
Time Frame: Measured from treatment initiation through Week 60
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 0.0 [0.0 to 30.8] | 0.0 [0.0 to 30.8]

27. Secondary Outcome: Percentage of Participants Who Had at Least One Serious Adverse Event Assessed as Related to Study Drug Through Week 60
Description: as for outcome 8
Time Frame: Measured from treatment initiation through Week 60
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 30.8]

28. Secondary Outcome: Percentage of Participants Who Had at Least One Adverse Event Assessed as Related to Study Drug That Led to Permanent Discontinuation of Study Drug Through Week 60
Description: as for outcome 5
Time Frame: Measured from treatment initiation through Week 60
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants | 0.0 [0.0 to 36.9] | 0.0 [0.0 to 28.5] | 0.0 [0.0 to 21.8] | 10.0 [0.3 to 44.5] | 0.0 [0.0 to 30.8]

29. Secondary Outcome: Percentage of Participants Who Experienced Virologic Failure Through Week 48
Description: Percentage of participants who experienced virologic failure based on the following definition: ART-experienced participants who had two subsequent viral loads greater or equal to 200 copies/mL at any time, or for ART-naive participants, two subsequent viral loads greater to or equal to 200 copies/mL at 24 weeks or after. The results are presented by ART experienced, ART naïve, and overall.
Time Frame: Measured from treatment initiation through Week 48
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants
  Overall | 12.5 | 0.0 | 0.0 | 0.0 | 0.0
  ART-experienced: number analyzed (Participants) | 5 | 11 | 15 | 10 | 10
  ART-experienced | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  ART-naive: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  ART-naive | 33.3 |  |  |  |

30. Secondary Outcome: Percentage of Participants Who Experienced Virologic Failure Through Week 60
Description: as for outcome 29
Time Frame: Measured from treatment initiation through Week 60
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants
  Overall | 12.5 | 0.0 | 0.0 | 0.0 | 0.0
  ART-experienced: number analyzed (Participants) | 5 | 11 | 15 | 10 | 10
  ART-experienced | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  ART-naive: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  ART-naive | 33.3 |  |  |  |

31. Secondary Outcome: Percentage of Participants With HIV-1 RNA Less Than 200 Copies/mL
Description: Viral loads less than the lower limit of quantification were imputed as one less than the lower limit.
Time Frame: Weeks 4, 24, and 48
Population: All participants taking treatment at timepoint who started treatment for their enrollment weight band and whose dose may have been increased to a higher weight band due to weight gain, who either completed treatment through Week 24 or discontinued treatment due to toxicity prior to Week 24. One participant in Weight Band #4 discontinued study treatment between Weeks 24 and 48, so this participant was excluded from analysis at Week 48.
Measure: Number; unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of participants
  Week 4 | 75.0 | 100.0 | 100.0 | 100.0 | 100.0
  Week 24 | 87.5 | 100.0 | 100.0 | 100.0 | 100.0
  Week 48: number analyzed (Participants) | 8 | 11 | 15 | 9 | 10
  Week 48 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0

32. Secondary Outcome: Percentage of Participants With Virologic Success of HIV-1 RNA Less Than 200 Copies/mL Using FDA Snapshot Algorithm
Description: Percentage of participants with virologic success of HIV-1 RNA less than 200 copies/mL using FDA snapshot algorithm at Weeks 4, 24, and 48. Viral loads less than the lower limit of quantification were imputed as one less than the lower limit.
Time Frame: Weeks 4, 24, and 48
Population: All participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 9 | 12 | 15 | 10 | 11
percentage of participants
  Week 4 | 66.7 [29.9 to 92.5] | 100.0 [73.5 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [71.5 to 100.0]
  Week 24 | 77.8 [40.0 to 97.2] | 91.7 [61.5 to 99.8] | 100.0 [78.2 to 100.0] | 100.0 [69.2 to 100.0] | 100.0 [71.5 to 100.0]
  Week 48 | 88.9 [51.8 to 99.7] | 91.7 [61.5 to 99.8] | 100.0 [78.2 to 100.0] | 90.0 [55.5 to 99.7] | 100.0 [71.5 to 100.0]

33. Secondary Outcome: Percentage of Participants With Virologic Success of HIV-1 RNA Less Than 50 Copies/mL Using FDA Snapshot Algorithm
Description: Percentage of participants with virologic success of HIV-1 RNA less than 50 copies/mL using FDA snapshot algorithm at Weeks 4, 24, and 48. Viral loads less than the lower limit of quantification were imputed as one less than the lower limit.
Time Frame: Weeks 4, 24, and 48
Population: All participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 9 | 12 | 15 | 10 | 11
percentage of participants
  Week 4 | 44.4 [13.7 to 78.8] | 91.7 [61.5 to 99.8] | 86.7 [59.5 to 98.3] | 80.0 [44.4 to 97.5] | 100.0 [71.5 to 100.0]
  Week 24 | 77.8 [40.0 to 97.2] | 83.3 [51.6 to 97.9] | 93.3 [68.1 to 99.8] | 100.0 [69.2 to 100.0] | 100.0 [71.5 to 100.0]
  Week 48 | 77.8 [40.0 to 97.2] | 66.7 [34.9 to 90.1] | 86.7 [59.5 to 98.3] | 70.0 [34.8 to 93.3] | 90.9 [58.7 to 99.8]

34. Secondary Outcome: Median (Q1, Q3) CD4+ Cell Count
Description: Per protocol, CD4 + cell counts were not required at Week 60. CD4 results were therefore analyzed through Week 48. For participants who discontinued study drug prior to the other timepoints due to safety or virologic failure, results imputed using the baseline value.
Time Frame: Weeks 4, 24, and 48
Population: All participants taking treatment at timepoint who started treatment for their enrollment weight band and whose dose may have been increased to a higher weight band due to weight gain, who either completed treatment through Week 24 or discontinued treatment due to toxicity prior to Week 24.
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
cells/mm^3
  Week 4 | 3528 [1458 to 4457] | 1385 [1020 to 1761] | 812 [716 to 1164] | 992 [930 to 1408] | 841 [627 to 1238]
  Week 24 | 2208 [1302 to 2939] | 1184 [987 to 1810] | 894 [689 to 1250] | 944 [774 to 1047] | 920 [675 to 1188]
  Week 48 | 1853 [1287 to 2700] | 1235 [889 to 1591] | 930 [791 to 1274] | 942 [765 to 1194] | 777 [681 to 825]

35. Secondary Outcome: Median (Q1, Q3) CD4+ Percentage
Description: Per protocol, CD4+ cell count percentages were not required at Week 60. CD4 results were therefore analyzed through Week 48. For participants who discontinued study drug prior to the other timepoints due to safety or virologic failure, results imputed using the baseline value.
Time Frame: Weeks 4, 24, and 48
Population: as for outcome 34
Measure: Median (Inter-Quartile Range); unit: percentage of CD4+ in total lymphocytes
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
percentage of CD4+ in total lymphocytes
  Week 4 | 41.6 [31.4 to 43.6] | 33.9 [30.2 to 39.5] | 32.4 [27.8 to 39.7] | 34.4 [30.0 to 41.0] | 39.5 [38.2 to 41.0]
  Week 24 | 36.6 [29.3 to 40.3] | 35.2 [27.3 to 40.0] | 33.5 [25.9 to 40.1] | 37.7 [27.0 to 42.0] | 38.6 [36.0 to 44.1]
  Week 48 | 34.8 [29.5 to 42.6] | 34.1 [26.7 to 39.9] | 30.5 [29.3 to 41.0] | 33.5 [28.5 to 37.0] | 37.6 [34.0 to 41.4]

36. Secondary Outcome: Median (Q1,Q3) Change From Baseline in Total Cholesterol
Description: Baseline is defined as the latest pre-dose assessment with a non-missing value. Where time was not collected, assessments on the day of treatment initiation are assumed to be taken prior to first dose. Missing results for participants who discontinued study treatment prior to the specified timepoint due to safety or virologic failure were imputed using the baseline value. Per protocol, there was no expectation of evaluating lipids in a fasting state for this study. A relative few participants were identified as having been in a fasted state at a given study visit, but the majority did not fast for this evaluation.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 34
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
mmol/L
  Baseline to Week 24 | -0.31 [-0.84 to 0.68] | -0.70 [-1.40 to 0.49] | -0.67 [-0.94 to 0.16] | -0.32 [-0.65 to 0.34] | -0.18 [-0.67 to 0.10]
  Baseline to Week 48 | 0.00 [-0.84 to 0.67] | -0.50 [-1.30 to 0.01] | -0.68 [-1.10 to -0.39] | -0.25 [-0.73 to 0.23] | -0.09 [-0.39 to 0.13]

37. Secondary Outcome: Median (Q1,Q3) Change From Baseline in HDL
Description: as for outcome 36
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 34
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
mmol/L
  Baseline to Week 24 | -0.01 [-0.21 to 0.24] | -0.06 [-0.40 to 0.10] | -0.19 [-0.30 to 0.00] | -0.15 [-0.40 to 0.20] | -0.06 [-0.18 to 0.16]
  Baseline to Week 48 | -0.10 [-0.26 to 0.18] | -0.20 [-0.30 to 0.10] | -0.24 [-0.37 to -0.08] | -0.19 [-0.50 to 0.33] | 0.05 [-0.01 to 0.13]

38. Secondary Outcome: Median (Q1,Q3) Change From Baseline in LDL
Description: as for outcome 36
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 34
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
mmol/L
  Baseline to Week 24 | 0.18 [-0.78 to 0.52] | -0.20 [-0.70 to 0.31] | -0.26 [-0.70 to 0.11] | -0.22 [-0.60 to 0.25] | -0.21 [-0.73 to -0.03]
  Baseline to Week 48 | 0.05 [-0.52 to 1.14] | -0.13 [-1.20 to 0.42] | -0.30 [-0.60 to 0.10] | 0.00 [-0.18 to 0.13] | 0.03 [-0.41 to 0.50]

39. Secondary Outcome: Median (Q1,Q3) Change From Baseline in Triglycerides
Description: as for outcome 36
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 34
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 10
mmol/L
  Baseline to Week 24 | -0.51 [-1.28 to 0.06] | -0.51 [-0.80 to -0.13] | -0.17 [-0.58 to 0.32] | -0.20 [-0.38 to 0.16] | -0.24 [-0.73 to 0.89]
  Baseline to Week 48 | -0.43 [-0.97 to 0.07] | -0.32 [-0.90 to 0.30] | -0.21 [-0.60 to 0.20] | 0.00 [-0.31 to 0.10] | -0.27 [-1.27 to -0.01]

40. Secondary Outcome: Parent/Guardian-reported Percent Adherence to Study Drug
Description: Parent/guardian-reported percent adherence to study drug in the 30 days prior to the study visit according to adherence questionnaire responses.
Time Frame: Weeks 4, 24, and 48
Population: All participants taking treatment at timepoint who received at least one dose of study treatment. One participant in Weight Band #4 discontinued treatment following the Week 24 visit and was not included in analysis at Week 48.
Measure: Median (Full Range); unit: percentage of study drug taken
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
percentage of study drug taken
  Week 4 | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [97.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [95.0 to 100.0]
  Week 24 | 100.0 [100.0 to 100.0] | 100.0 [95.0 to 100.0] | 100.0 [90.0 to 100.0] | 100.0 [90.0 to 100.0] | 100.0 [95.0 to 100.0]
  Week 48: number analyzed (Participants) | 8 | 11 | 15 | 9 | 11
  Week 48 | 100.0 [60.0 to 100.0] | 100.0 [90.0 to 100.0] | 100.0 [85.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [99.0 to 100.0]

41. Secondary Outcome: Parent/Guardian-reported Number of Missed Doses of Study Drug
Description: Parent/guardian-reported number of missed doses of study drug in the 30 days prior to the study visit according to adherence questionnaire responses.
Time Frame: Weeks 4, 24, and 48
Population: as for outcome 40
Measure: Median (Full Range); unit: missed doses
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
missed doses
  Week 4 | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 1] | 0 [0 to 0] | 0 [0 to 1]
  Week 24 | 0 [0 to 0] | 0 [0 to 1] | 0 [0 to 2] | 0 [0 to 0] | 0 [0 to 0]
  Week 48: number analyzed (Participants) | 8 | 11 | 15 | 9 | 11
  Week 48 | 0 [0 to 5] | 0 [0 to 6] | 0 [0 to 5] | 0 [0 to 0] | 0 [0 to 1]

42. Secondary Outcome: Parent/Guardian-reported Reason for Missed Doses of Study Drug
Description: Parent/guardian-reported reason for missed doses of study drug in the 30 days prior to the study visit according to adherence questionnaire responses.
Time Frame: Weeks 4, 24, and 48
Population: All participants taking treatment at timepoint who received at least one dose of study treatment. One participant in Weight Band #4 discontinued treatment following the Week 24 visit and was not included in analysis at Week 48. All other instances of missing data were due to participants with no missed doses not responding to this question specifying the reason.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
Participants
  Week 4: number analyzed (Participants) | 8 | 10 | 15 | 10 | 11
  Week 4: Both parents were admitted in the hospital | 0 | 0 | 0 | 0 | 0
  Week 4: Caregiver too sick | 0 | 0 | 0 | 0 | 0
  Week 4: Caregiver was too busy to give the medication | 0 | 0 | 0 | 0 | 0
  Week 4: Change in daily routine | 0 | 0 | 0 | 0 | 0
  Week 4: Forgot to administer medication | 0 | 0 | 1 | 0 | 0
  Week 4: Mom was in a hurry and forgot to give child medication | 0 | 0 | 0 | 0 | 1
  Week 4: Tried to spit it out because of taste (away from caregiver) | 0 | 0 | 0 | 0 | 0
  Week 4: No missed doses | 8 | 10 | 14 | 10 | 10
  Week 24: number analyzed (Participants) | 7 | 10 | 14 | 10 | 10
  Week 24: Both parents were admitted in the hospital | 0 | 0 | 0 | 0 | 0
  Week 24: Caregiver too sick | 0 | 0 | 1 | 0 | 0
  Week 24: Caregiver was too busy to give the medication | 0 | 0 | 0 | 0 | 0
  Week 24: Change in daily routine | 0 | 1 | 0 | 0 | 0
  Week 24: Forgot to administer medication | 0 | 1 | 0 | 0 | 0
  Week 24: Mom was in a hurry and forgot to give child medication | 0 | 0 | 0 | 0 | 0
  Week 24: Tried to spit it out because of taste (away from caregiver) | 0 | 0 | 0 | 1 | 0
  Week 24: No missed doses | 7 | 8 | 13 | 9 | 10
  Week 48: number analyzed (Participants) | 7 | 11 | 15 | 9 | 11
  Week 48: Both parents were admitted in the hospital | 1 | 0 | 0 | 0 | 0
  Week 48: Caregiver too sick | 0 | 0 | 0 | 0 | 0
  Week 48: Caregiver was too busy to give the medication | 1 | 0 | 0 | 0 | 0
  Week 48: Change in daily routine | 0 | 1 | 0 | 0 | 1
  Week 48: Forgot to administer medication | 0 | 1 | 1 | 0 | 0
  Week 48: Mom was in a hurry and forgot to give child medication | 0 | 0 | 0 | 0 | 0
  Week 48: Tried to spit it out because of taste (away from caregiver) | 0 | 0 | 0 | 0 | 0
  Week 48: No missed doses | 5 | 9 | 14 | 9 | 10

43. Secondary Outcome: Parent/Guardian-reported Response of How Well the Person Usually Responsible Administered the Study Drug in the Way They Were Supposed to
Description: Parent/guardian-reported response of how well the person usually responsible administered the study drug in the way they were supposed to in the 30 days prior to the study visit according to adherence questionnaire responses.
Time Frame: Weeks 4, 24, and 48
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
Participants
  Week 4: Excellent | 4 | 7 | 12 | 7 | 9
  Week 4: Very good | 3 | 4 | 2 | 2 | 2
  Week 4: Good | 1 | 0 | 1 | 1 | 0
  Week 4: Fair | 0 | 0 | 0 | 0 | 0
  Week 4: Poor | 0 | 0 | 0 | 0 | 0
  Week 24: Excellent | 2 | 7 | 10 | 5 | 9
  Week 24: Very good | 5 | 3 | 4 | 1 | 2
  Week 24: Good | 1 | 1 | 1 | 3 | 0
  Week 24: Fair | 0 | 0 | 0 | 0 | 0
  Week 24: Poor | 0 | 0 | 0 | 1 | 0
  Week 48: number analyzed (Participants) | 8 | 11 | 15 | 9 | 11
  Week 48: Excellent | 2 | 7 | 12 | 7 | 11
  Week 48: Very good | 5 | 3 | 2 | 1 | 0
  Week 48: Good | 0 | 1 | 1 | 1 | 0
  Week 48: Fair | 1 | 0 | 0 | 0 | 0
  Week 48: Poor | 0 | 0 | 0 | 0 | 0

44. Secondary Outcome: Parent/Guardian-reported Response of How Often the Child Received the Study Drug in the Way They Were Supposed to
Description: Parent/guardian-reported response of how often the child received the study drug in the way they were supposed to in the 30 days prior to the study visit according to adherence questionnaire responses.
Time Frame: Weeks 4, 24, and 48
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
Participants
  Week 4: Always | 8 | 9 | 14 | 10 | 10
  Week 4: Almost always | 0 | 0 | 1 | 0 | 1
  Week 4: Usually | 0 | 1 | 0 | 0 | 0
  Week 4: Sometimes | 0 | 0 | 0 | 0 | 0
  Week 4: Never | 0 | 1 | 0 | 0 | 0
  Week 24: Always | 7 | 9 | 12 | 6 | 9
  Week 24: Almost always | 1 | 2 | 3 | 2 | 2
  Week 24: Usually | 0 | 0 | 0 | 1 | 0
  Week 24: Sometimes | 0 | 0 | 0 | 0 | 0
  Week 24: Never | 0 | 0 | 0 | 1 | 0
  Week 48: number analyzed (Participants) | 8 | 11 | 15 | 9 | 11
  Week 48: Always | 6 | 7 | 13 | 9 | 11
  Week 48: Almost always | 0 | 3 | 1 | 0 | 0
  Week 48: Usually | 1 | 0 | 1 | 0 | 0
  Week 48: Sometimes | 1 | 0 | 0 | 0 | 0
  Week 48: Never | 0 | 1 | 0 | 0 | 0

45. Secondary Outcome: Parent/Guardian-reported Ease of Giving Study Drug
Description: Parent/guardian-reported ease of giving study drug according to palatability questionnaire responses.
Time Frame: Weeks 4, 12, 24, and 48
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
Participants
  Week 4: The child takes by themselves easily | 0 | 2 | 11 | 9 | 9
  Week 4: The child takes easily with help | 6 | 8 | 4 | 0 | 2
  Week 4: The child takes with help but you need to threaten, bribe, or promise a reward | 0 | 1 | 0 | 1 | 0
  Week 4: You need to hold and force the child | 2 | 0 | 0 | 0 | 0
  Week 12: The child takes by themselves easily | 0 | 5 | 10 | 7 | 9
  Week 12: The child takes easily with help | 8 | 5 | 5 | 2 | 2
  Week 12: The child takes with help but you need to threaten, bribe, or promise a reward | 0 | 1 | 0 | 1 | 0
  Week 12: You need to hold and force the child | 0 | 0 | 0 | 0 | 0
  Week 24: The child takes by themselves easily | 0 | 3 | 12 | 8 | 8
  Week 24: The child takes easily with help | 8 | 6 | 3 | 2 | 3
  Week 24: The child takes with help but you need to threaten, bribe, or promise a reward | 0 | 2 | 0 | 0 | 0
  Week 24: You need to hold and force the child | 0 | 0 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 8 | 11 | 15 | 9 | 11
  Week 48: The child takes by themselves easily | 0 | 4 | 10 | 6 | 10
  Week 48: The child takes easily with help | 8 | 5 | 4 | 2 | 1
  Week 48: The child takes with help but you need to threaten, bribe, or promise a reward | 0 | 1 | 1 | 1 | 0
  Week 48: You need to hold and force the child | 0 | 1 | 0 | 0 | 0

46. Secondary Outcome: Parent/Guardian-reported Response of Child's Face When Taking Study Drug
Description: Parent/guardian-reported response of child's face when taking study drug according to palatability questionnaire responses.
Time Frame: Weeks 4, 12, 24, and 48
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
Participants
  Week 4: Very good | 1 | 5 | 0 | 2 | 5
  Week 4: Good | 1 | 4 | 10 | 2 | 2
  Week 4: Average | 4 | 2 | 4 | 3 | 4
  Week 4: Bad | 1 | 0 | 1 | 2 | 0
  Week 4: Very bad | 1 | 0 | 0 | 1 | 0
  Week 12: Very good | 2 | 3 | 4 | 3 | 6
  Week 12: Good | 2 | 3 | 5 | 3 | 2
  Week 12: Average | 4 | 4 | 3 | 2 | 3
  Week 12: Bad | 0 | 0 | 2 | 1 | 0
  Week 12: Very bad | 0 | 1 | 1 | 1 | 0
  Week 24: Very good | 2 | 5 | 5 | 3 | 6
  Week 24: Good | 3 | 3 | 4 | 2 | 4
  Week 24: Average | 2 | 3 | 3 | 3 | 1
  Week 24: Bad | 1 | 0 | 2 | 2 | 0
  Week 24: Very bad | 0 | 0 | 1 | 0 | 0
  Week 48: number analyzed (Participants) | 8 | 11 | 15 | 9 | 11
  Week 48: Very good | 3 | 5 | 5 | 3 | 6
  Week 48: Good | 2 | 4 | 6 | 3 | 0
  Week 48: Average | 3 | 1 | 1 | 1 | 5
  Week 48: Bad | 0 | 0 | 1 | 1 | 0
  Week 48: Very bad | 0 | 1 | 2 | 1 | 0

47. Secondary Outcome: Parent/Guardian-reported Response of Child's Face When Taking Favorite Food
Description: Parent/guardian-reported response of child's face when taking favorite food according to palatability questionnaire responses.
Time Frame: Weeks 4, 12, 24, and 48
Population: as for outcome 40
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 11
Participants
  Week 4: Very good | 3 | 7 | 4 | 4 | 8
  Week 4: Good | 4 | 3 | 9 | 3 | 2
  Week 4: Average | 1 | 1 | 2 | 3 | 1
  Week 4: Bad | 0 | 0 | 0 | 0 | 0
  Week 4: Very bad | 0 | 0 | 0 | 0 | 0
  Week 12: Very good | 4 | 6 | 7 | 6 | 10
  Week 12: Good | 1 | 2 | 4 | 3 | 1
  Week 12: Average | 3 | 3 | 3 | 0 | 0
  Week 12: Bad | 0 | 0 | 0 | 1 | 0
  Week 12: Very bad | 0 | 0 | 1 | 0 | 0
  Week 24: Very good | 6 | 6 | 8 | 6 | 10
  Week 24: Good | 1 | 4 | 5 | 2 | 0
  Week 24: Average | 1 | 1 | 2 | 1 | 1
  Week 24: Bad | 0 | 0 | 0 | 1 | 0
  Week 24: Very bad | 0 | 0 | 0 | 0 | 0
  Week 48: number analyzed (Participants) | 8 | 11 | 15 | 9 | 11
  Week 48: Very good | 8 | 7 | 9 | 7 | 11
  Week 48: Good | 0 | 4 | 6 | 2 | 0
  Week 48: Average | 0 | 0 | 0 | 0 | 0
  Week 48: Bad | 0 | 0 | 0 | 0 | 0
  Week 48: Very bad | 0 | 0 | 0 | 0 | 0

48. Secondary Outcome: Parent/Guardian-reported Time for Study Drug Tablets to Dissolve
Description: Parent/guardian-reported time for study drug tablets to dissolve according to acceptability questionnaire responses
Time Frame: Weeks 4, 12, 24, and 48
Population: All participants taking treatment at timepoint who received at least one dose of study treatment. One participant in Weight Band #4 prematurely discontinued treatment and was not included in analysis at Week 48. Weight Band #5 dosing was not in tablet form, so this question did not apply to Weight Band #5 or to Weight Band #4 participants following dose escalation.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 0
Participants
  Week 4: Less than 1 minute | 3 | 5 | 0 | 2 |
  Week 4: 1 to less than 3 minutes | 3 | 5 | 11 | 7 |
  Week 4: 3 to 5 minutes | 2 | 1 | 4 | 1 |
  Week 12: Less than 1 minute | 2 | 2 | 4 | 1 |
  Week 12: 1 to less than 3 minutes | 5 | 7 | 8 | 6 |
  Week 12: 3 to 5 minutes | 1 | 2 | 3 | 3 |
  Week 24: Less than 1 minute | 2 | 5 | 4 | 3 |
  Week 24: 1 to less than 3 minutes | 5 | 6 | 10 | 5 |
  Week 24: 3 to 5 minutes | 1 | 0 | 1 | 2 |
  Week 48: number analyzed (Participants) | 8 | 11 | 15 | 4 | 0
  Week 48: Less than 1 minute | 3 | 4 | 2 | 2 |
  Week 48: 1 to less than 3 minutes | 3 | 6 | 11 | 2 |
  Week 48: 3 to 5 minutes | 2 | 1 | 2 | 0 |

49. Secondary Outcome: Parent/Guardian-reported Satisfaction With the Number of Study Drug Tablets to Dissolve
Description: Parent/guardian-reported satisfaction with the number of study drug tablets to dissolve according to acceptability questionnaire responses
Time Frame: Weeks 4, 12, 24, and 48
Population: as for outcome 48
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 8 | 11 | 15 | 10 | 0
Participants
  Week 4: It is acceptable | 7 | 10 | 15 | 8 |
  Week 4: It is too many | 1 | 1 | 0 | 2 |
  Week 4: It is too few | 0 | 0 | 0 | 0 |
  Week 12: It is acceptable | 8 | 11 | 15 | 9 |
  Week 12: It is too many | 0 | 0 | 0 | 1 |
  Week 12: It is too few | 0 | 0 | 0 | 0 |
  Week 24: It is acceptable | 8 | 10 | 14 | 10 |
  Week 24: It is too many | 0 | 1 | 1 | 0 |
  Week 24: It is too few | 0 | 0 | 0 | 0 |
  Week 48: number analyzed (Participants) | 8 | 11 | 15 | 4 | 0
  Week 48: It is acceptable | 7 | 11 | 15 | 4 |
  Week 48: It is too many | 0 | 0 | 0 | 0 |
  Week 48: It is too few | 1 | 0 | 0 | 0 |

50. Secondary Outcome: Antiretroviral (ARV) Resistance Mutations
Description: ARV resistance mutations at time of virologic failure and at entry for children with virologic failure.
Time Frame: Entry and confirmation of virologic failure
Population: Participants experiencing confirmed virologic failure. Due to assay limitations, mutation results could not be obtained from the specimen collected at the virologic failure confirmation visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0
Participants
  Entry Visit: Integrase K14R | 1 |  |  |  |
  Entry Visit: Integrase A21T | 1 |  |  |  |
  Entry Visit: Integrase V31I | 1 |  |  |  |
  Entry Visit: Integrase V72I | 1 |  |  |  |
  Entry Visit: Integrase L74I | 1 |  |  |  |
  Entry Visit: Integrase T112V | 1 |  |  |  |
  Entry Visit: Integrase V113I | 1 |  |  |  |
  Entry Visit: Integrase T125A | 1 |  |  |  |
  Entry Visit: Integrase V126L | 1 |  |  |  |
  Entry Visit: Integrase G134N | 1 |  |  |  |
  Entry Visit: Integrase I135V | 1 |  |  |  |
  Entry Visit: Integrase K136R | 1 |  |  |  |
  Entry Visit: Integrase V165I | 1 |  |  |  |
  Entry Visit: Integrase A196P | 1 |  |  |  |
  Entry Visit: Integrase V236I | 1 |  |  |  |
  Entry Visit: Integrase V281M | 1 |  |  |  |
  Entry Visit: Integrase S283G | 1 |  |  |  |
  Entry Visit: Protease L10V | 1 |  |  |  |
  Entry Visit: Protease I13V | 1 |  |  |  |
  Entry Visit: Protease G16E | 1 |  |  |  |
  Entry Visit: Protease E35D | 1 |  |  |  |
  Entry Visit: Protease M36I | 1 |  |  |  |
  Entry Visit: Protease R41K | 1 |  |  |  |
  Entry Visit: Protease K43R | 1 |  |  |  |
  Entry Visit: Protease H69K | 1 |  |  |  |
  Entry Visit: Protease I72V | 1 |  |  |  |
  Entry Visit: Protease L89M | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase E6D | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase K11T | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase K20R | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase V35T | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase T39K | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase K43E | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase Q102K | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase K122E | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase D123S | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase C162S | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase T165I | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase K173A | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase Q174K | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase D177E | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase T200A | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase I202V | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase Q207A | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase L210M | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase R211S | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase V245E | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase A272P | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase R277K | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase T286A | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase L295L/I | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase E312N | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase I326V | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase I329V | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase G335D | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase M357K | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase K358R | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase G359S | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase K366R | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase A371V | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase T377S | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase K390R | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase K395R | 1 |  |  |  |
  Entry Visit: Reverse Transcriptase A400T | 1 |  |  |  |

ADVERSE EVENTS:
Time Frame: From study entry to study completion (at Week 48 or 60) or premature study discontinuation
Description: All adverse events (i.e., all grade 1 or higher) identified after enrollment were collected and entered into adverse event electronic case report forms (eCRFs). For any event involving a hypersensitivity reaction to ABC, additional data was also collected and entered into other designated eCRFs
  The definition of the term adverse event provided in Version 2.0 of the DAIDS EAE Manual was used in this study
Arm/Group | Weight Band #1 (6 to Less Than 10 kg at Study Entry) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) | Weight Band #5 (25 kg or Greater at Study Entry)
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12 | 0/15 | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/9 | 1/12 | 0/15 | 1/10 | 0/11
Other Adverse Events (participants affected / at risk) | 8/9 | 10/12 | 15/15 | 10/10 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Weight Band #1 (6 to Less Than 10 kg at Study Entry) (N=9) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) (N=12) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) (N=15) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) (N=10) | Weight Band #5 (25 kg or Greater at Study Entry) (N=11)
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Weight Band #1 (6 to Less Than 10 kg at Study Entry) (N=9) | Weight Band #2 (10 to Less Than 14 kg at Study Entry) (N=12) | Weight Band #3 (14 to Less Than 20 kg at Study Entry) (N=15) | Weight Band #4 (20 to Less Than 25 kg at Study Entry) (N=10) | Weight Band #5 (25 kg or Greater at Study Entry) (N=11)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 0 | 3
Secondary thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Otorrhoea (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Conjunctival pallor (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gingival swelling (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Facial pain (General disorders) | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 2 | 2 | 1 | 0
Swelling face (General disorders) | 0 | 0 | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 1 | 0 | 1 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 3 | 1 | 0
Otitis media chronic (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tinea capitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tinea faciei (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Adverse event following immunisation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 3 | 8 | 7 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 5 | 4 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 2 | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 3 | 3 | 2
Blood creatinine increased (Investigations) | 4 | 6 | 6 | 5 | 5
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood pressure systolic increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 3 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 6 | 5 | 9 | 9 | 7
Haemoglobin decreased (Investigations) | 2 | 0 | 0 | 1 | 1
Low density lipoprotein increased (Investigations) | 1 | 0 | 1 | 2 | 1
Neutrophil count decreased (Investigations) | 1 | 1 | 2 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0
Underweight (Metabolism and nutrition disorders) | 2 | 0 | 4 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 0
Nightmare (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Childhood asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 5 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1 | 0
Nasal flaring (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 3 | 1 | 2
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Tonsillar exudate (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-08-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT03760458/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/58/NCT03760458/SAP_001.pdf